CLINICAL TRIAL: NCT00000708
Title: Multi-center Comparison of Fluconazole (UK-49,858) and Amphotericin B as Treatment for Acute Cryptococcal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 059; Protocol 159; Project 056; Investigator 556
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1991-07

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Injections, Intravenous; Cryptococcus neoformans; Cryptococcosis; Drug Therapy, Combination; Fluconazole; Administration, Oral; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Flucytosine; Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Flucytosine
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To compare the safety and effectiveness of fluconazole (FCZ) and amphotericin B (AMB), alone or in combination with flucytosine (FLC), as treatment for acute cryptococcal meningitis in patients who have not been treated previously or who have relapsed after a previous successful treatment.

Cryptococcal meningitis is an important cause of disease and death among patients with AIDS. Usually AMB is given either alone or with FLC to patients with this infection, but these treatments are not always effective and both have toxic effects. Animal studies and preliminary studies in humans show that FCZ is active in cryptococcal meningitis and suggest that it may be less toxic than either AMB or FLC.

DETAILED DESCRIPTION:
Cryptococcal meningitis is an important cause of disease and death among patients with AIDS. Usually AMB is given either alone or with FLC to patients with this infection, but these treatments are not always effective and both have toxic effects. Animal studies and preliminary studies in humans show that FCZ is active in cryptococcal meningitis and suggest that it may be less toxic than either AMB or FLC.

Patients accepted into the study are randomly assigned to FCZ or AMB. Patients assigned to FCZ take FCZ by mouth daily for 10 weeks. Patients assigned to AMB are given intravenous injections of AMB daily for 6-10 weeks. Non-AIDS patients assigned to AMB also take FLC by mouth daily. The use of FLC in patients with AIDS is decided on an individual basis. Patients with AIDS who respond satisfactorily to FCZ receive maintenance therapy to prevent relapse for an additional 12 months. Patients with AIDS who respond to AMB may qualify for another Pfizer Central Research protocol. Patients without AIDS who respond to therapy are observed for 6 months for relapse. During therapy, samples of blood and cerebrospinal fluid (by lumbar puncture) are taken periodically in order to evaluate the effectiveness of the drug treatments and to identify possible toxic effects.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Immunosuppressant therapy.
* Cyclosporin plasma concentrations should be monitored and appropriate dosage adjustments made when used with amphotericin B or fluconazole.
* Antiviral therapy.
* Prophylaxis for Pneumocystis carinii pneumonia.
* Treatment of intercurrent opportunistic infection as long as no investigational agent, or approved agent for an investigational indication, is used.
* Antipyretics, hydrocortisone, or meperidine to prevent or ameliorate side effects associated with amphotericin B.

Concurrent Treatment:

Allowed:

- Radiation therapy for mucocutaneous Kaposi's sarcoma.

Patients must have:

* Written informed consent obtained from the patient or from the patient's legal guardian.
* One of the following:
* (1) Tentative identification of Cryptococcus neoformans in culture of lumbar cerebrospinal fluid (CSF). Results of baseline cultures need not be available when therapy is begun, but therapy is discontinued if the baseline CSF culture is later found to be negative for C. neoformans, or (2) Clinical and CSF findings (cell count, protein, glucose) compatible with cryptococcal meningitis plus one of the following:
* (a) Positive CSF India ink examination, (b) Culture or biopsy evidence of extraneural cryptococcal infection, (c) Positive serum of CSF cryptococcal antigen test, or increase in titer for previously treated patients with suspected relapse, or (d) Biopsy evidence of central nervous system cryptococcal infection.
* Treatment status of either no prior systemic antifungal therapy for cryptococcosis or relapse after prior therapy. The success of prior therapy must have been documented by negative CSF culture at the end of therapy.

Prior Medication:

Allowed within 4 weeks of study entry:

- Successful prior therapy for cryptococcosis, but no more than 1 mg/kg/week amphotericin B.

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy.
* Prophylaxis for Pneumocystis carinii pneumonia.

Exclusion Criteria

Co-existing Condition:

Excluded:

* Acute or chronic meningitis based on any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles, or amphotericin B.
* Moderate or severe liver disease defined as any one or more of the following:
* SGOT or SGPT > 5 x upper limit of normal, total bilirubin > 2.5 mg/dl, prothrombin time > 5 seconds over control, or alkaline phosphatase > 2 x upper limit of normal.
* Comatose patients.

Concurrent Medication:

Excluded:

* Drugs with low therapeutic ratios that undergo hepatic metabolism may not be used with fluconazole until possible drug interactions have been clarified.
* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.
* Systemic antifungal agent other than the assigned study drug.

Concurrent Treatment:

Excluded:

Lymphocyte replacement.

Prior Medication:

Excluded within 4 weeks of study entry:

* More than 1 mg/kg/week amphotericin B.

Patients unlikely to survive more than 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Primary Completion 1991-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armstrong D, Study Chair
Locations (6):
- United States (6):
  - Univ of Miami School of Medicine, Miami, Florida
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Powderly WG. Recent advances in the management of cryptococcal meningitis in patients with AIDS. Clin Infect Dis. 1996 May;22 Suppl 2:S119-23. doi: 10.1093/clinids/22.supplement_2.s119. PMID 8722838
- [Background] Powderly WG, Cloud GA, Dismukes WE, Saag MS. Measurement of cryptococcal antigen in serum and cerebrospinal fluid: value in the management of AIDS-associated cryptococcal meningitis. Clin Infect Dis. 1994 May;18(5):789-92. doi: 10.1093/clinids/18.5.789. PMID 8075272
- [Background] Saag MS, Powderly WG, Cloud GA, Robinson P, Grieco MH, Sharkey PK, Thompson SE, Sugar AM, Tuazon CU, Fisher JF, et al. Comparison of amphotericin B with fluconazole in the treatment of acute AIDS-associated cryptococcal meningitis. The NIAID Mycoses Study Group and the AIDS Clinical Trials Group. N Engl J Med. 1992 Jan 9;326(2):83-9. doi: 10.1056/NEJM199201093260202. PMID 1727236